CLINICAL TRIAL: NCT04037202
Title: Effect of Foot Massage on Postpartum Comfort and Pain Level of the Mothers Who Had Vaginal Birth: A Randomised Controlled Trial
Brief Title: Effect of Foot Massage on Postpartum Comfort and Pain Level of the Mothers Who Had Vaginal Birth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Rabia Genç, Associate Professor, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0000-0002-6762-0496
Record Dates: First submitted 2019-07-24; First posted 2019-07-30 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Postpartum Disorder; Massage
Keywords: analgesia; massage; midwifery; pain; postpartum period
MeSH Terms: conditions — Puerperal Disorders; Agnosia; Pain

STUDY DESIGN:
Intervention Model Description: The researcher prepared the mother for foot massage (foot care, proper position, etc.) and gave a total of 20-minute massage of foot massage, 10 minutes for each foot. VAS was repeated immediately after the first session (in the 20th minute) and after 30 minutes (in the 50th minute). The second session was performed on the second day, 20-24 hours after the first session (before the discharge). The VAS was analyzed before the second (last) session (0th minute), and the VAS was repeated immediately after the application (20th minute) and 30 minutes (50th minute), and the PCS was administered for the last time. Administered analgesics were recorded in the DFC and the administration made with package leaflet was supported.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): The first session of the foot massage was performed after mothers were taken to the postpartum service and after the effect of the first analgesia had elapsed (4-6 hours after birth).
  The researcher prepared the mother for foot massage (foot care, proper position, etc.) and gave a total of 20-minute massage of foot massage, 10 minutes for each foot. VAS was repeated immediately after the first session (in the 20th minute) and after 30 minutes (in the 50th minute). The second session was performed on the second day, 20-24 hours after the first session (before the discharge). The VAS was analyzed before the second (last) session (0th minute), and the VAS was repeated immediately after the application (20th minute) and 30 minutes (50th minute), and the PCS was administered for the last time. Administered analgesics were recorded in the DFC and the administration made with package leaflet was supported.
  Interventions: Other: Foot massage
- Control Group (No Intervention): Routine procedures were applied and VAS was repeated at the same time periodical as the study group mothers (0th, 20th and 50th minute) and after 20-24 hours (before discharge), at the same time intervals (0th, 20th and 50th minute) pain status was measured by using VAS and PCS was administered for the last time and analgesics administered were recorded on the DFC.

INTERVENTIONS:
Other: Foot massage — Foot massage includes classical massage techniques such as effleurage, petrissage and friction techniques. Effleurage is the movement of stroking and lubricating superficial tissues. Therefore, it is performed at the beginning and ending of the massage. Petrissage is the slow and rhythmic movement to apply direct pressure to the soft tissue underlying the skin with the balls of the fingers and thumbs. Friction is the application of pressure through small circular movements only in small areas, using hand or fingers. While muscle tissue is compressed and relaxed, blood and lymph circulation increases. Thus, lactic acid in the muscle fibers is diminished and fatigue and stress are decreased.
  Arms: Study Group

SUMMARY:
Background and Purpose: This study aims to investigate the effect of foot massage in the postpartum period on the need of receiving analgesic medication after assessing the postpartum comfort and pain status of the mothers who had vaginal delivery.Materials and methods: The study was completed with 66 mothers. As data collection tools, a questionnaire, Postpartum Comfort Scale (PCS), Visual Analogue Scale (VAS) and Drug Follow-up Card (DFC) were used.

DETAILED DESCRIPTION:
Background and purpose: This study aims to investigate the effect of foot massage in the postpartum period on the need of receiving analgesic medication after assessing the postpartum comfort and pain status of the mothers who had vaginal delivery.

Materials and methods: In order to keep the number of people in balance between the groups, "block randomization" method which is one of the fixed probability randomization types was preferred. The research was completed with 66 persons, 33 in the study group and 33 in the control group. As data collection tools, a questionnaire, Postpartum Comfort Scale (PCS), Visual Analogue Scale (VAS) and Drug Follow-up Card (DFC) were used.

Research inclusion criteria include (i) primipara mothers (who had their first birth), (ii) mothers who had normal vaginal delivery, (iii) those who had undergone episiotomy, (iv) who were volunteered to participate in the study, (v) who were on the first day of delivery (first 24 hours), (vi) who had no complications in the infant and the baby, (vii) age of whom ranged from 18 to 35, (viii) those who did not apply or receive any other complementary therapy, (ix) mothers who did not have any wound, infection or discomfort etc. on their feet, and those who can read and write.

ELIGIBILITY:
Inclusion Criteria:

* primipara mothers (who had their first birth),
* mothers who had normal vaginal delivery,
* those who had undergone episiotomy,
* who were volunteered to participate in the study,
* who were on the first day of delivery (first 24 hours),
* who had no complications in the infant and the baby,
* age of whom ranged from 18 to 35,
* those who did not apply or receive any other complementary therapy,
* mothers who did not have any wound, infection or discomfort etc. on their feet,
* mothers who can read and write

Exclusion Criteria:

* mothers with any systemic disease
* mothers who dislike foot massage during practice
* early discharge mothers
* mothers who applied another massage technique
* mothers who take the analgesic drug unnecessarily

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Informed Consent Form | 5-10 minutes
  The form consists of 31 questions about family, pregnancy, birth and newborn characteristics.This form was completed during the first meeting at the hospital.
Postpartum Comfort Scale (PCS) | 5-10 minutes
  In accordance with the comfort theory developed by Katharine Kolcaba in 1994, the PCS developed by Karakaplan and Yıldız (2010) consists of 34 items.A 5-point Likert-type scoring system was used to evaluate each item.Expression and scoring were made for each item ranging from "totally agree" (5 points), and "strongly disagree" (1 points).In positive sentences, "I fully agree" indicates the best comfort (5 points) and in negative sentences low comfort (1 points).Accordingly, the lowest score to be taken from the scale is 34 and the highest score is 170.
Visual Analog Scale (VAS) | Less than 1 minute
  It is a single-item continuous scale consisting of a horizontal or vertical line and is usually 10 centimeters (100 mm) in length. For example, the severity of pain a patient feels ranges from "no pain" with 0 points on a line to "severe pain" with 10 points.Scoring is achieved by measuring the point the patient has marked with a ruler.Pain relief points in VAS;
  * Absence of pain (0-4 mm),
  * Slight pain (5-44 mm),
  * Moderate pain (45-74 mm)
  * Severe pain (75-100 mm)
Drug Follow-up Card (DFC) | About 1 minute
  The researcher was prepared, this is a follow-up card in which the name and surname of the mothers, the name of the drug given to the mothers, the route of administration of the drug, date / time and dosage are indicated.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Izmir, Bornova, Turkey (Türkiye)

REFERENCES:
- [Background] Simavli S, Kaygusuz I, Gumus I, Usluogullari B, Yildirim M, Kafali H. Effect of music therapy during vaginal delivery on postpartum pain relief and mental health. J Affect Disord. 2014 Mar;156:194-9. doi: 10.1016/j.jad.2013.12.027. Epub 2013 Dec 28. PMID 24411681
- [Background] Abbaspoor Z, Akbari M, Najar S. Effect of foot and hand massage in post-cesarean section pain control: a randomized control trial. Pain Manag Nurs. 2014 Mar;15(1):132-6. doi: 10.1016/j.pmn.2012.07.008. Epub 2013 Jan 24. PMID 23352729
- [Background] Saatsaz S, Rezaei R, Alipour A, Beheshti Z. Massage as adjuvant therapy in the management of post-cesarean pain and anxiety: A randomized clinical trial. Complement Ther Clin Pract. 2016 Aug;24:92-8. doi: 10.1016/j.ctcp.2016.05.014. Epub 2016 May 30. PMID 27502807
- [Background] Asazawa K PhD, Kato Y Bs, Yamaguchi A Ms, Inoue A Bs. The Effect of Aromatherapy Treatment on Fatigue and Relaxation for Mothers during the Early Puerperal Period in Japan: A Pilot Study. Int J Community Based Nurs Midwifery. 2017 Oct;5(4):365-375. PMID 29043282
- [Background] Xue M, Fan L, Ge LN, Zhang Y, Ge JL, Gu J, Wang Y, Chen Y. Postoperative Foot Massage for Patients after Caesarean Delivery. Z Geburtshilfe Neonatol. 2016 Aug;220(4):173-8. doi: 10.1055/s-0042-104802. Epub 2016 Aug 10. PMID 27509141
- [Background] Degirmen N, Ozerdogan N, Sayiner D, Kosgeroglu N, Ayranci U. Effectiveness of foot and hand massage in postcesarean pain control in a group of Turkish pregnant women. Appl Nurs Res. 2010 Aug;23(3):153-8. doi: 10.1016/j.apnr.2008.08.001. Epub 2009 Jan 15. PMID 20643325
- [Background] Eogan M, Daly L, O'Herlihy C. The effect of regular antenatal perineal massage on postnatal pain and anal sphincter injury: a prospective observational study. J Matern Fetal Neonatal Med. 2006 Apr;19(4):225-9. doi: 10.1080/14767050600593155. PMID 16854696
- [Background] Wang HL, Keck JF. Foot and hand massage as an intervention for postoperative pain. Pain Manag Nurs. 2004 Jun;5(2):59-65. doi: 10.1016/j.pmn.2004.01.002. PMID 15297952
- [Background] Coban A, Sirin A. Effect of foot massage to decrease physiological lower leg oedema in late pregnancy: a randomized controlled trial in Turkey. Int J Nurs Pract. 2010 Oct;16(5):454-60. doi: 10.1111/j.1440-172X.2010.01869.x. PMID 20854342
- [Background] Santos Jde O, Oliveira SM, Nobre MR, Aranha AC, Alvarenga MB. A randomised clinical trial of the effect of low-level laser therapy for perineal pain and healing after episiotomy: a pilot study. Midwifery. 2012 Oct;28(5):e653-9. doi: 10.1016/j.midw.2011.07.009. Epub 2011 Oct 5. PMID 21982202
- [Background] Aksoy Derya Y, Pasinlioglu T. The Effect of Nursing Care Based on Comfort Theory on Women's Postpartum Comfort Levels After Caesarean Sections. Int J Nurs Knowl. 2017 Jul;28(3):138-144. doi: 10.1111/2047-3095.12122. Epub 2015 Nov 25. PMID 26602188
- [Background] Senol DK, Aslan E. The Effects of Cold Application to the Perineum on Pain Relief After Vaginal Birth. Asian Nurs Res (Korean Soc Nurs Sci). 2017 Dec;11(4):276-282. doi: 10.1016/j.anr.2017.11.001. Epub 2017 Nov 26. PMID 29290275
- [Background] Moghimi-Hanjani S, Mehdizadeh-Tourzani Z, Shoghi M. The Effect of Foot Reflexology on Anxiety, Pain, and Outcomes of the Labor in Primigravida Women. Acta Med Iran. 2015 Aug;53(8):507-11. PMID 26545996
- [Background] Jahdi F, Mehrabadi M, Mortazavi F, Haghani H. The Effect of Slow-Stroke Back Massage on the Anxiety Levels of Iranian Women on the First Postpartum Day. Iran Red Crescent Med J. 2016 Jun 7;18(8):e34270. doi: 10.5812/ircmj.34270. eCollection 2016 Aug. PMID 27781122
- [Background] Adib-Hajbaghery M, Abasi A, Rajabi-Beheshtabad R. Whole body massage for reducing anxiety and stabilizing vital signs of patients in cardiac care unit. Med J Islam Repub Iran. 2014 Jun 17;28:47. eCollection 2014. PMID 25405113
- [Background] Can HO, Saruhan A. Evaluation of the effects of ice massage applied to large intestine 4 (hegu) on postpartum pain during the active phase of labor. Iran J Nurs Midwifery Res. 2015 Jan-Feb;20(1):129-38. PMID 25709702
- [Background] Hattan J, King L, Griffiths P. The impact of foot massage and guided relaxation following cardiac surgery: a randomized controlled trial. J Adv Nurs. 2002 Jan;37(2):199-207. doi: 10.1046/j.1365-2648.2002.02083.x. PMID 11851788
- [Derived] Deussen AR, Ashwood P, Martis R, Stewart F, Grzeskowiak LE. Relief of pain due to uterine cramping/involution after birth. Cochrane Database Syst Rev. 2020 Oct 20;10(10):CD004908. doi: 10.1002/14651858.CD004908.pub3. PMID 33078388
- See also: Factors that affecting mothers' postnatal comfort — http://www.diclemedj.org/upload/sayi/20/Dicle%20Med%20J-01507.pdf
- See also: Effect of Uterine Massage in the Perception of Women's Postpartum Pain Intensity — https://dergipark.org.tr/download/article-file/205618